CLINICAL TRIAL: NCT05756959
Title: Myopia Control Combined PBM With Myopic Defocus Lens in Children: Double-blind RCT for 6 Month
Brief Title: Myopia Control Combined PBM With Myopic Defocus Lens in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Collaborators: The First People's Hospital of Xuzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Xuzhou First People's Hospital
Record Dates: First submitted 2023-02-05; First posted 2023-03-07 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PBM therapy + SVS (Experimental): Low lever red light therapy with single vision spectacles
  Interventions: Device: PBM; Device: Single vision spectacles
- Peripheral defocus spectacles (Experimental): a spectacles with special design with peripheral myopic defocus to control myopia progression
  Interventions: Device: Peripheral defocus spectacles
- PBM +Peripheral defocus spectacles (Experimental): Low lever red light therapy with a spectacles with special design with peripheral myopic defocus to control myopia progression
  Interventions: Device: PBM; Device: Peripheral defocus spectacles
- Control (Placebo Comparator): single vision spectacles only as the control
  Interventions: Device: Single vision spectacles

INTERVENTIONS:
Device: PBM — PBM, is a low intensity red light at wavelength of 650nm; Peripheral defocus spectacels is a peripheral design glasseses for correct myopia and control myopia
  Other Names: Low lever light therapy; low intensity red light therapy; low lever laser therapy; repeated red light therapy
  Arms: PBM +Peripheral defocus spectacles; PBM therapy + SVS
Device: Peripheral defocus spectacles — plus power design of many peripheral small lenses to achieve myopic defocus of the retina in the peripheral retina
  Other Names: Myopic defocus spectacles for myopia control
  Arms: PBM +Peripheral defocus spectacles; Peripheral defocus spectacles
Device: Single vision spectacles — Distance vision correction with the single vision spectacles for the myopia correction methods (glasseses for myopia correction)
  Other Names: single vision glasseses for myopia correction lenses
  Arms: Control; PBM therapy + SVS

SUMMARY:
To study the efficacy of myopi control with two methods: low lever red light and peripheral defocus spectacles with four groups and design with prospective, double-blind, randimized, and with control for 6 month.

DETAILED DESCRIPTION:
myopic children with age from 6 ~13 years old. And refraction from -0.50D~-5.50D.

The red light is low lever laser therapy at wavelength of 650nm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the supervision of the children
* 6~13 years old (including both the 6 and 13)
* SE range: -0.50~-5.50D
* Astigmatism <=2.00D
* BCVA >=0.8
* Anisometropia <=1.50D
* Confirmed to no use of other myopia control intervention

Exclusion Criteria:

* Ocular lesions to effect vision or diseases (such as cataract, glaucoma, marcular pathology, cornea lesions, uveitis, retina detachment, congential opitc abnormal and etc.)
* Halo, glare, toutic, ADHD, psoriasis
* Systom disease: immune disease, central nerve system, Down syndrome, asthma, severe cardiopulmonary abnormal, severe liver and renal dysfunction.
* Squint, ocular lesion or acute imflammation.
* Other myopia control interventions within recent 3 month such as atropine, device, orthokeratology, multi-focus soft lens, multi-function spectacles.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
axial length (mm) | 6 month
  Axial length changes at follow-up of 6 month from baseline will be measured by IOLmaster 500 at the same site by the same examiner with the mean values of 5 times measurements at either time.
  Changes in axial length (mm) without cycloplegia are to be measured by IOLmaster(Carl Zeiss). Five measurements will be taken and then averaged.
SE (Diopter, D) | 6 month
  changes of cycloplegic spherical equivalent from baseline will be measured under cycloplegic refraction by autorefractor. Five measured by the same autorefractor are to be obtained for each eye.

SECONDARY OUTCOMES:
UCVA (logMar visual acuity record) | 6 month
  Uncorrected visual acuity will be measured under 5-meter distance logMar Visual acuity chart without any aid （including the spectacles or contact lens) at baseline and at follow-up
BCVA (logMar visual acuity record) | 6 month
  Best corrected visual acuity will be measured under the same 5-meter distance logMar Visual acuity as the UCVA both at baseline and at follow-up.
OCT | 6-month
  Opitcal coherence tomography(OCT) record
  The marcular sturcture and image scanned by the optical coherent topography will be measured by linear scan at the marcular by the same Optical coherence tomography with the same examiner and the same instrument both at baseline and at follow-up
SFCT （um) | 6-month
  Sub-forveal choroidal thickness will be measured with the same software in the same Optical coherence tomography (OCT) at the location from the foveal center manually

OTHER OUTCOMES:
Adverse Event | 6 month
  Any adverse event reported by subjects or doctors related or un-related to the product during the whole study period

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, BA, Study Director — The First People's Hospital of Xuzhou
Locations (1):
- the first people's hospital of Xuzhou, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided